CLINICAL TRIAL: NCT01853098
Title: Effect of a Novel Mindfulness Based Loving Kindness Meditation on Positive and Negative Affect
Brief Title: A Pilot Study of Positive Affect Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Stefan G. Hofmann, Dr., Boston University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3151
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Affect (Mental Function); Compassion
Keywords: loving-kindness meditation; mindfulness meditation; compassion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Positive Affect Training (PAT) (Experimental): The intervention will be conducted in groups with 6-8 participants and 2 facilitators/therapists per group. The groups will meet once a week for 12 successive weeks and each session will be approximately 60 minutes long.
  Interventions: Behavioral: Positive Affect Training (PAT)

INTERVENTIONS:
Behavioral: Positive Affect Training (PAT) — During the PAT sessions, the participants will be taught the basics of mindfulness and how to concentrate their thoughts and feelings on the present moment in a non-judgmental fashion. As the therapy sessions continue, participants will be introduced to basic loving-kindness meditation (LKM). They will be taught to identify and focus the positive feelings they have when they are around someone or something they care about, and transfer these feelings first to themselves, then to a close friend, to a neutral individual, to people whom they dislike, and finally to all living beings.

SUMMARY:
The primary objective of this study is a proof-of-concept study to test whether a novel mindfulness based intervention, Positive Affect Training (PAT), can enhance positive affect and compassion, and decrease negative affect and feelings of depression. PAT involves a combination of practicing mindfulness meditation and loving-kindness meditation in groups. The goal of the research is to test the initial feasibility and efficacy in increasing positive affect and decreasing negative affect in individuals recruited from the general community who experience negative affect. If the training proves to be successful, we will test the intervention, in additional studies, on individuals with dysthymic disorder and other clinical disorders. PAT is a cost-effective, non-invasive intervention. Therefore if effective, it could be an alternative or supplemental intervention option to existing psychotherapy for dysthymic disorder.

DETAILED DESCRIPTION:
Loving-kindness meditation (LKM) and mindfulness meditation, in which PAT is rooted, are derived from Buddhist practices that have been empirically shown to have applications in improving mental health. Throughout the 1990s and early 2000s, mindfulness based CBT was shown to decrease stress, negative affect, and chronic pain in both psychiatric and non-psychiatric subjects. Mindfulness-based therapy has since been shown to be effective for treating mood and anxiety disorders. Only recently has LKM been examined as an intervention for affective symptoms. This meditation practice seems to be particularly suited for reducing negative affect while also enhancing positive affect in individuals who show emotional dysregulation, such as people with dysthymic disorder. This notion is supported by experimental studies suggesting that LKM decreases anxiety and stress, positively influences emotional responses to neutral stimuli, and promotes positive emotions such as trust, love, hope, and compassion. Dr. Fredrickson, a prominent researcher and social psychologist who is the foremost expert in LKM will serve as an outside consultant for the development of the protocol. She is not listed as an official collaborator because she will not be in direct contact with the participant data that the investigators will collect.

The intervention the investigators plan to develop, Positive Affect Training (PAT), combines mindfulness and LKM, with a strong emphasis on the latter. The investigators will adopt strategies that have been described in a previous LKM protocol for trauma victims. The investigators contacted Dr. Kearney who shared his manual with us. Given the impressive effect LKM seems to have on generating positive, and attenuating negative affect in experimental studies, the investigators plan to test PAT as a method of improving positive affect. The current study aims to test the initial efficacy of PAT in individuals who report experiencing a low mood. The investigators hypothesize significant improvement in subjects' self-reported ratings of negative and positive affect as a result of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Responds positively to the question on the recruitment material (flyer and posting): "Have you been feeling depressed or in a low mood for most of the day, more days than not, nearly every day for 1 year or longer?"
* Must have a negative affect scale score of the PANAS of at least 21.6 (1 SD above the mean of normative sample)

Exclusion Criteria:

* Participants with a BDI score of 30 or higher (more than moderate depression) will be excluded.
* Participants who are at risk of harming themselves will be excluded from participating in the study. Suicidality will be assessed after obtaining consent during the screening visit. In addition, the Beck Depression Inventory will be examined for self-reported suidicality. If a participant is found to have suicidal ideation, the PI will be contacted immediately and appropriate follow-up care will be provided by referring the participant to the ER.
* Participants will be assessed through a phone screen using questions from the Anxiety Disorders Interview Schedule (ADIS) for disorders that could impose a safety risk for the participants or others (e.g., bipolar disorder, schizophrenia, etc). Subjects who endorse "yes" responses to phone screen items will be excluded.
* Participants who are receiving any psychiatric or psychological treatment for a mood or anxiety disorder at the time of the assessment will be excluded from the study. Participants who initiate such treatments while being enrolled in the study will be closely monitored. These participants will be allowed to remain in the study, but will later be excluded from the data analyses. They are allowed to remain in the study for ethical reasons and because the present trial is a proof-of-concept study and not a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Positive and Negative Affect Scale (PANAS) | 12 weeks

SECONDARY OUTCOMES:
Change from Baseline in Self-Compassion Scale (SCS) | 12 weeks
Change from Baseline in Beck Anxiety and Depression Scale (BDI) | 12 weeks
Change from Baseline in Compassionate Love Scale | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stefan G. Hofmann, Ph.D., Principal Investigator — Boston University, Psychology Department
Locations (1):
- Center for Anxiety and Related Disorders at Boston University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028
- [Background] Hofmann SG, Sawyer AT, Fang A, Asnaani A. Emotion dysregulation model of mood and anxiety disorders. Depress Anxiety. 2012 May;29(5):409-16. doi: 10.1002/da.21888. Epub 2012 Mar 16. PMID 22430982
- [Background] Hofmann SG, Grossman P, Hinton DE. Loving-kindness and compassion meditation: potential for psychological interventions. Clin Psychol Rev. 2011 Nov;31(7):1126-32. doi: 10.1016/j.cpr.2011.07.003. Epub 2011 Jul 26. PMID 21840289
- [Background] Carson JW, Keefe FJ, Lynch TR, Carson KM, Goli V, Fras AM, Thorp SR. Loving-kindness meditation for chronic low back pain: results from a pilot trial. J Holist Nurs. 2005 Sep;23(3):287-304. doi: 10.1177/0898010105277651. PMID 16049118
- [Background] Hutcherson CA, Seppala EM, Gross JJ. Loving-kindness meditation increases social connectedness. Emotion. 2008 Oct;8(5):720-4. doi: 10.1037/a0013237. PMID 18837623
- [Background] Fredrickson BL, Cohn MA, Coffey KA, Pek J, Finkel SM. Open hearts build lives: positive emotions, induced through loving-kindness meditation, build consequential personal resources. J Pers Soc Psychol. 2008 Nov;95(5):1045-1062. doi: 10.1037/a0013262. PMID 18954193
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865